CLINICAL TRIAL: NCT04372680
Title: WeanINg From Mechanical Ventilation for ARDS CovId-19 Patients Guided by Combined Thoracic UltraSound: a Prospective, Multicenter, Randomized, Open-label, Parallel-group Clinical Trial
Brief Title: WeanINg From Mechanical Ventilation for ARDS CovId-19 Patients Guided by Combined Thoracic UltraSound.
Acronym: INVICTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/20/0138; 2020-A00916-33 (Other: ID-RCB)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; ARDS, Human; Mechanical Ventilation
Keywords: COVID-19,; ARDS; Mechanical ventilation; Lung ultrasound; Echocardiography
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Controlled, open-label, in parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTUS strategy group (Experimental): CTUS examination will be performed until the day of patient extubation. CTUS examination will consist on a fully bedside ultrasonographic assessment of lung, cardiac and diaphragm functions
  Interventions: Diagnostic Test: CTUS examination
- standard strategy group (No Intervention): from the day of patient's inclusion and beyond every day, the clinical team in charge of patients will decide to perform or not an SBT following current recommendations2. These criteria are mainly based on clinical data and do not include any specific ultrasound assessment.

INTERVENTIONS:
Diagnostic Test: CTUS examination — fully bedside ultrasonographic assessment of lung, cardiac and diaphragm functions
  Arms: CTUS strategy group

SUMMARY:
The most feared complication of COVID-19 infection is the occurrence of an acute respiratory distress syndrome (ARDS) that requires ICU admission and prolonged mechanical ventilation in more than 2% of the affected patients. Establishing the correct time to extubate mechanically ventilated patients is a crucial issue in the critical care practice. Delayed extubation has several consequences such as patient's mortality, health-care-related complications, neuropsychological adverse events. The aim of the INVICTUS study is to evaluate whether a CTUS-based MV weaning strategy could reduce the duration of mechanical ventilation of ARDS COVID-19 ICU patients by 72 hours, compared with usual medical care.

DETAILED DESCRIPTION:
Identifying patients at risk for postextubation distress using standard clinical criteria and the only available test the investigators have, that is, the spontaneous breathing trial (SBT) remains a challenging issue2. A cumulative body of evidence suggest that the decision to attempt extubation might be assisted by the use of thoracic ultrasound. This non-invasive, reproducible and fully bedside approach is able to provide accurate information about respiratory, cardiac and neuromuscular functions which are independent predictors of extubation outcome. Recently, the investigators have demonstrated that a combined thoracic ultrasound (CTUS) strategy based on lung ultrasound, echocardiography and diaphragm ultrasonographic assessment data performs better than routine clinical assessment to evaluate extubation readiness in medical and surgical ICU patients3. CTUS appears as a unique point of care precision medicine prognostic and diagnostic tool for the management of patients experiencing ARDS. Based on those premises, the investigators hypothesize that CTUS-based MV weaning strategy could reduce the duration of mechanical ventilation of ARDS COVID-19 ICU patients by 72 hours, compared with usual medical care. This research is a national, multicenter, randomized, controlled, open-label, in parallel group. Patients will be randomized on 1:1 CTUS strategy group or standard strategy group, daily daily followed until extubation+48hours, reassessed at day 28 and at 3 months. In CTUS strategy group, a combined CTUS examination will be performed until the day of patient extubation. CTUS examination will consist on a fully bedside ultrasonographic assessment of lung, cardiac and diaphragm functions. In standard strategy group, from the day of patient's inclusion and beyond every day, the clinical team in charge of patients will decide to perform or not an SBT following current recommendations2. These criteria are mainly based on clinical data and do not include any specific ultrasound assessment.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission for severe acute respiratory distress syndrome (ARDS, as previously defined5 by a ratio of the partial pressure of arterial oxygen to the fraction of inspired oxygen of less than 150) related to COVID-19.
* Non paralyzed because of neuromuscular blocking agents.
* Ventilated patient in pressure support mode for at least 6 hours and at most 24 hours.
* Surrogate decision maker's consent.
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* Reduction or cessation of active treatment.
* Paraplegia with medullar level more than T8.
* Tracheostomy before hospital admission.
* History of severe respiratory illness.
* Patient under juridical protection.
* Pregnancy or nursing woman.
* Enrolled in another trial evaluating mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Delay from the start of Mechanical Ventilation weaning process to extubation | day 28
  Delay from the start of MV weaning process (day of the switch from volume control mode to pressure support ventilation) to extubation (or spontaneously breathing through tracheostomy cannula) for at least 48 hours, as previously defined.

SECONDARY OUTCOMES:
delay from intubation to extubation | day 28
  delay from intubation to extubation
Successful of extubation | day 28
  Successful of extubation if patient is not reintubated after 48 hours of extubation
mortality rate | day 28
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice RIU-POULENC, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU de LIMOGES, Limoges
  - CHU de TOULOUSE, Toulouse

IPD SHARING:
Plan to Share IPD: No